CLINICAL TRIAL: NCT02337244
Title: Persona Outcomes Led Assessment Research in Total Knee Arthroplasty (POLAR - TKA)
Brief Title: Zimmer POLAR Persona - TKA (EMEA Study)
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer, GmbH (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: CSE2013-07K
Record Dates: First submitted 2015-01-06; First posted 2015-01-13 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Severe Knee Pain; Severe Knee Disability; Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Polyarthritis
Keywords: Osteoarthritis; Rheumatoid arthritis; Traumatic arthritis; Polyarthritis; Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Zimmer Persona Total Knee System — No Intervention
  Other Names: Primary Knee Replacement; Total Knee Arthroplasty; Total Knee Replacement

SUMMARY:
The primary objective of this study is to obtain implant survivorship and clinical outcomes data for commercially available Persona knee implants used in primary total knee arthroplasty. The assessment will include:

1. Implant survivorship based on removal of a study device.
2. Safety based on incidence and frequency of adverse events.
3. Clinical performance measured by overall pain and function, quality of life data, radiographic parameters and survivorship.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-controlled study of the commercially available Persona knee implants. The study will require each site to obtain Ethics approval prior to study enrollment. All potential study subjects will be required to participate in the Informed Consent Process.

Study subjects will undergo preoperative clinical evaluations prior to their total knee arthroplasty. The post-operative clinical and radiographic evaluations will be conducted at 5 days to 6 weeks, 3 to 6 months, 1 year, 2, 3, 4, and 5 years after implantation. The hospital CHU Clermont-Ferrand, France with PI Prof. Boisgard will conduct additional 7 (voluntary) and 10 years (standard of care) follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18-75 years of age, inclusive.
* Patient qualifies for primary total knee arthroplasty based on physical exam and medical history, including diagnosis of severe knee pain and disability due to at least one of the following:

  * rheumatoid arthritis, osteoarthritis, traumatic arthritis, polyarthritis;
  * collagen disorders and/or avascular necrosis of the femoral condyle;
  * post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy;
  * moderate valgus, varus, or flexion deformities;
  * the salvage of previously failed surgical attempts that did not include partial or total knee arthroplasty of the ipsilateral knee.
* Patient is willing and able to complete scheduled study procedures and follow-up evaluations.
* Independent of study participation, patient is a candidate for commercially available Zimmer Persona knee implants implanted in accordance with product labeling.

Exclusion Criteria:

* Patient is currently participating in any other surgical intervention studies or pain management studies.
* Previous history of infection in the affected joint and/or other local/systemic infection that may affect the prosthetic joint.
* Insufficient bone stock on femoral or tibial surfaces.
* Skeletal immaturity.
* Neuropathic arthropathy.
* Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb.
* Stable, painless arthrodesis in a satisfactory functional position.
* Severe instability secondary to the absence of collateral ligament integrity.
* Rheumatoid arthritis accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin.
* Patient has a known or suspected sensitivity or allergy to one or more of the implant materials.
* Patient is pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.).
* Patient has previously received partial or total knee arthroplasty for the ipsilateral knee.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary total knee arthroplasty subjects that receive the Zimmer Persona Total Knee System.
Sampling Method: Non-Probability Sample
Enrollment: 777 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Kaplan-Meier Implant Survivorship | 5 years
  Kaplan-Meier survivorship at 5 years with revision of any implant component, for any reason, as endpoint.

SECONDARY OUTCOMES:
'Knee injury and Osteoarthritis Outcome Score' (KOOS) subscale scores. | 5 years
  The scores related to the five KOOS subscales calculated at different time points until 5 years.
'Forgotten Joint Score' (FJS-12) | 5 years
  The score related to the FJS-12 patient-reported questionaire calculated at different time points until 5 years.
Oxford Knee Score (OKS) | 5 years
  The score related to the OKS patient-reported questionaire calculated at different time points until 5 years.
EuroQol (EQ)-5D-3L score and EQ 'Visual Analog Scale' (VAS) | 5 years
  The scores related to the EQ-5D-3L questionnaire and the EQ-VAS calculated at different time points until 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dominkus, MD, Principal Investigator — Orthopädisches Spital Speising, Wien, Austria; Hendrik Verburg, MD, Principal Investigator — Stichting Research Orthopedie & Reinier de Graaf Groep, Delf, Netherlands; Nicholas London, MD, Principal Investigator — Harrogate and District NHS, Harrogate, England; Stéphane Boisgard, MD, Principal Investigator — CHU de Clermont-Ferrand, Clermont-Ferrand, France; François Canovas, Prof, Principal Investigator — Hospital Lapeyronie, Montpellier; Pere Torner, MD, Principal Investigator — Hospital Parc Tauli, Sabadell; Jon Clarke, MD, Principal Investigator — Golden Jubilee National Hospital, Clydebank; David Deehan, Prof, Principal Investigator — Freeman Hospital, Newcastle; Karl Dieter Heller, Prof, Principal Investigator — HEH Braunschweig; Fritz Thorey, Prof, Principal Investigator — Atos Klinik Heidelberg; Fernando Martinez Delgado, MD, Principal Investigator — Hospital Miguel Servet Zaragoza; Hermant Pandit, Prof, Principal Investigator — University of Leeds
Locations (12):
- Orthopädisches Spital Speising, Vienna, Austria
- France (2):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier régional Universitaire de Montpellier, Montpellier
- Germany (2):
  - HEH Braunschweig, Braunschweig
  - Atos Klinik Heidelberg, Heidelberg
- Stichting Research Orthopedie & Reinier de Graaf Groep, Delft, Netherlands
- Spain (2):
  - Hospital Parc Tauli, Sabadell
  - Hospital Miguel Servet, Zaragoza
- United Kingdom (4):
  - University of Leeds, Leeds, Leeds/UK
  - Golden Jubilee National Hospital, Clydebank
  - Harrogate and District NHS, Harrogate
  - The Newcastle Upon Tyne Hospitals, Newcastle

REFERENCES:
- [Derived] Mathijssen NMC, Verburg H, London NJ, Landsiedl M, Dominkus M. Patient reported outcomes and implant survivorship after Total knee arthroplasty with the persona knee implant system: two year follow up. BMC Musculoskelet Disord. 2019 Mar 4;20(1):97. doi: 10.1186/s12891-019-2470-y. PMID 30832636